CLINICAL TRIAL: NCT00339703
Title: Levels of Serum Resistin in Asthmatics as a Potential Marker of Systemic Inflammation and Disease State.
Status: Completed | Type: Observational
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Principal Investigator, Capt Jeffrey LaRochelle, USAF, MC, Physician, 59th Medical Wing
Other Study IDs: FWH20040210H
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Asthma
Keywords: Resistin; Asthma; CRP; Diabetes; FIZZ
MeSH Terms: conditions — Asthma; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Subjects between the ages of 18 and 65 without a diagnosis of asthma or other inflammatory disease were enrolled from the patient population at Wilford Hall Medical Center. Subjects underwent a single blood draw and spirometer.
- Mild to Moderate Asthma: Subjects between the ages of 18 and 65, who were previously diagnosed with moderate to severe persistent asthma as defined by the National Asthma Education and Prevention Program (NAEPP), were enrolled from the Allergy and Immunology clinic at Wilford Hall Medical Center. Subjects on inhaled corticosteroids or other controller medications were allowed in the study, but subjects on oral corticosteroids were excluded. Subjects underwent a single blood draw and spirometer.

SUMMARY:
The purpose of this study is to determine whether serum resistin levels in asthmatics are elevated. We will recruit subjects from the allergy/immunology clinic with a prior diagnosis of moderate to severe persistent asthma in addition to subjects being seen for evaluation of drug allergies. Based on the inclusion and exclusion criteria below, subjects will be placed into a control and asthma group. Each subject will undergo one blood draw in the main lab at WHMC, and return a lavender top tube to the allergy/immunology clinic for the EIA resistin assay. The patient will then have a brief encounter with a physician to determine an up to date history of asthma symptoms prior to participating in the exhaled NO test. The entire subject encounter will take place with one clinic visit, and requires no follow up visits as part of the study. The greatest risk to each subject will be the blood draw, as the exhaled NO is a completely non-invasive test.

Plasma from each subject will be stored in a -70° freezer for no more than one month. Samples will be analyzed for resistin levels using an EIA assay run monthly. Mean values from serum CRP, serum glucose, serum resistin, and exhaled NO will be compared using a students T-test.

DETAILED DESCRIPTION:
Resistin is part of the FIZZ (found in inflammatory zones) family of genes, and was first characterized in murine models where it has been extensively studied as a potential link between type II diabetes and obesity. The murine FIZZ gene family consists of three related gene products: a)FIZZ-1 or Relm-a is found in adipocytes and lung tissue, b)FIZZ-2 or Relm-b found in the gastrointestinal tract, and c)FIZZ-3 or Resistin also found in adipocytes.1 Mouse models have shown resistin to be linked to obesity and insulin resistance, and thiazolidinedione has been shown to decrease resistin expression in mouse adipocytes.2 Distribution of the FIZZ gene products in humans is similar to mouse models: a)Relm-a is found in adipose, heart, and lung, b)Relm-b is found in the gastrointestinal tract, and c)Resistin is found in adipocytes and interestingly, is also found in circulating macrophages.3 Given the findings correlating obesity with diabetes in the mouse model, several studies were done in humans attempting to illustrate this same link. A study comparing middle age type II diabetics with matched controls found serum resistin levels to be increased in the diabetic group (16.6 vs 13.5, p<0.004), but this elevation was independent of adiposity, BMI, or insulin resistance. Elevation in C-reactive protein (CRP) in the diabetic group was the only factor that consistently correlated with elevation in resistin levels in this study.4 A second study comparing older (60-75 years of age) type II diabetics also found a significant elevation in serum resistin in the diabetic group that was independent of gender, insulin resistance, BMI, blood pressure, or total cholesterol. Interestingly, this study did find an association with plasma glucose concentration and serum resistin levels.5 Although there seems to be no direct link between resistin and insulin resistance in humans, the above data suggest a role for insulin in systemic inflammation commonly associated with diabetes. Adipocytes are known to be a source of inflammatory cytokines such as TNF-a and IL-6. TNF-a has been shown to be elevated in obesity, and many acute phase reactants and cytokines are associated with diabetes and the metabolic syndrome.6 In addition, resistin has been shown to induce VCAM-1, ICAM-1, and long pentraxin 3 (markers of vascular inflammation) in mouse models. The resistin related induction of VCAM-1 was partially blocked with a statin, indicating a role for resistin in vascular inflammation that may contribute to atherosclerosis and coronary artery disease seen in diabetics and the metabolic syndrome.7 Given the effects on vascular inflammation, resistin may be an important cytokine involved in a common inflammatory pathway seen in both diabetics and asthmatics.

Like diabetes, asthma is a disease marked by chronic inflammation. The inflammation associated with asthma has been predominantly illustrated in the airways, however, studies have shown that induced bronchoconstriction and asthma do illicit a systemic response with elevations in CRP thought to be mediated by IL-1, IL-6, and TNF-a via activated macrophages.8,9 In addition, CCL2 contributes to airway hyper-reactivity and cell migration, and thiazolidinedione has been shown to inhibit the IL-1b and TNF-a induced expression of CCL2 in the lung.10 Finally, a recent study illustrated an IL-4 and IL-13 induction of Relm-b via STAT-6 in response to allergic asthma.11 The level of serum resistin in human asthmatics is currently unknown, and may represent an important systemic marker of inflammation in this disease. Relating levels of serum resistin with disease state in conjunction with measurements of serum CRP and glucose would be an important aspect of further understanding the potential systemic inflammatory implications of asthma. In addition, unpublished data on exhaled NO have shown a positive correlation with asthma that could be used to further strengthen evidence of systemic inflammation with airway inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the asthmatic group will consist of the following: (a) male or non-pregnant female, (b) 18-65 years of age, (c) asthma defined as moderate or severe persistent by NHLBI guidelines, and characterized by at least daily symptoms, night symptoms at least once weekly, and a FEV1 between 60-80% of predicted. Newly diagnosed asthmatics, poorly controlled asthmatics, and hospitalized patients with asthma flares may also be considered in separate arms of this study.
* Inclusion criteria for the control group will consist of the following: (a) male or non-pregnant female, (b) 18-65 years of age.

Exclusion Criteria:

* Exlusion criteria for the asthmatic group will consist of the following: (a) current use of oral steroids or statins, (b) any serious concurrent disease process such as, but not limited to diabetes, coronary artery disease, or vasculitis, that would have effects on levels of systemic inflammation.
* Exclusion criteria for the control group will consist of the following: (a) current use of oral steroids or statins, (b) prior diagnosis of asthma, or clinical symptoms consistent with asthma or reactive airway disease, (c) any serious concurrent disease process such as, but not limited to diabetes, coronary artery disease, or vasculitis, that would have effects on levels of systemic inflammation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients enrolled to Wilford Hall Medical Center meeting the above eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2004-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S LaRochelle, MD, Principal Investigator — United States Air Force
Locations (1):
- Wilford Hall Medical Center, San Antonio, Texas, United States